CLINICAL TRIAL: NCT07184671
Title: Clinical, Radiological, Tissue and Biological Phenotyping for the Analysis of the Transition From Physiology to Pathology in Pulmonary Diseases With Pulmonary Hypertension.
Acronym: PHENOPULM
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00420-49
Record Dates: First submitted 2025-09-02; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Hypertension; Chronic Pulmonary Disease
Keywords: Pulmonary hypertension; chronic pulmonary disease; Phenotyping; Vascular remodeling
MeSH Terms: conditions — Hypertension, Pulmonary; Vascular Remodeling | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with chronic pulmonary disease and pulmonary hypertension: Patients on the lung transplant list with chronic pulmonary disease and pulmonary hypertension
  Interventions: Biological: blood sampling; Biological: broncho-alveolar lavage sampling; Biological: lung parenchyma sampling
- Control patients with chronic pulmonary disease without pulmonary hypertension: Control patients with chronic pulmonary disease without pulmonary hypertension on the lung transplant list or with an indication for lung resection surgery for diagnostic or therapeutic purposes.
  Interventions: Biological: blood sampling; Biological: broncho-alveolar lavage sampling; Biological: lung parenchyma sampling
- Control patients without chronic pulmonary disease or pulmonary hypertension: Control patients without chronic pulmonary disease or pulmonary hypertension with an indication for lung resection.
  Interventions: Biological: blood sampling; Biological: broncho-alveolar lavage sampling; Biological: lung parenchyma sampling

INTERVENTIONS:
Biological: blood sampling — 22mL peripheral blood will be collected
Biological: broncho-alveolar lavage sampling — Collected on resected tissue
Biological: lung parenchyma sampling — Collected on resected tissue

SUMMARY:
This is a monocentric, case-control, comparative study aiming at investigating the transition from physiological to pathological pulmonary circulation in patients with pulmonary hypertension (PH) and chronic lung diseases. The study will include 105 adults participants undergoing lung surgery, divided into three groups, Group A (patients with chronic lung disease and PH undergoing lung transplantation), Group B (patients with chronic lung disease without PH), and Group C (patients without chronic lung disease nor PH). The primary objective is to identify the association between vascular remodeling and PH by measuring the medial thickness of pulmonary arteries. Secondary objectives include multimodal phenotyping (clinical, radiological, tissue, and biological) to explore mechanisms of PH development. Blood, broncho-alveolar lavage, and lung tissue samples will be collected during routine care. The study aims to improve understanding of PH pathophysiology and identify potential biomarkers and therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years of age
2. Patient who has received information about the study and has not expressed any objection
3. Patient who is a beneficiary or entitled person under a social security scheme
4. Patient requiring thoracic surgery for an acute or chronic acquired pathology with planned resection of lung parenchyma.
5. Group A: patients on the lung transplant list with chronic lung disease and pulmonary hypertension*.

Group B: control patients with chronic lung disease without pulmonary hypertension on the lung transplant list or with an indication for lung resection surgery for diagnostic or therapeutic purposes.

Group C: control patients without chronic lung disease or pulmonary hypertension with an indication for lung resection.

*Pulmonary hypertension is defined by a mean resting pulmonary arterial pressure of 20 mmHg and pulmonary vascular resistances > 2UW and an occlusion pulmonary arterial pressure ≤ 15 mmHg.

Exclusion Criteria:

1. Person in exclusion period from another research protocol at the time the no-objection is collected
2. Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code (minors, adults under guardianship or trusteeship, patients deprived of their liberty, pregnant or breast-feeding women).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will be carried out on a continuous, daily basis in the thoracic surgery department of the Hôpital Nord in Marseille.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of pulmonary artery media thickness measured by optical microscopy | Surgical intervention

SECONDARY OUTCOMES:
Quantify endovascular (angiophagy) and perivascular (fibrosis, pro-inflammatory cells) tissue lesions. | Surgical intervention
  number of stage I, II and III angiophagia lesions relative to the number of arteries analyzed on a field of anatomopathology slides and classified according to artery diameter; surface area of pulmonary fibrosis relative to the total surface area of the tissue field explored; quantification of immune system cells in interstitial tissue relative to the tissue surface area explored.
Compare the radiological phenotyping of patients with pulmonary hypertension and without pulmonary hypertension, determined from patient lung scans | Baseline
Compare cardiorespiratory functional clinical phenotyping between patients with pulmonary hypertension and without pulmonary hypertension. | Baseline
  Using generalized linear model for assesment of respiratory function tests, 6-minute walk test and echocardiography of patients
Compare the biological phenotyping of biological lung inflammation from bronchioloalveolar lavage of patients with pulmonary hypertension and without pulmonary hypertension. | Surgical intervention
  Dosage of inflammatory proteins (IL1, IL10, IL6, etc.) and cytological analysis of bronchioloalveolar lavage
High-throughput proteomic quantification indices of circulating serum from patients with pulmonary hypertension compared with patients without pulmonary hypertension. | Baseline
Compare the phenotyping of pulmonary vascular microstructure by microCT in patients with pulmonary hypertension and without pulmonary hypertension. | Surgical intervention
Compare protein tissue phenotyping of pulmonary hypertension regulatory pathways in patients with and without pulmonary hypertension evaluated with Elisa tests on lung parenchyma. | Surgical intervention
Evaluate the statistical relationships between tissue vascular remodeling and tissue, alveolar, and blood protein alterations. | Baseline and surgical intervention
Compare genetic tissue phenotyping of pulmonary hypertension regulatory pathways in patients with and without pulmonary hypertension evaluated with PCR tests on lung parenchyma. | Surgical intervention